CLINICAL TRIAL: NCT06671873
Title: A Single-center, Open-label, Single-dose Phase I Clinical Study to Investigate the Human Mass Balance in Healthy Chinese Adult Male Subjects Following a Single Oral Dose of 250 mg/100 µCi [14C] HMPL-306
Brief Title: Study on Mass Balance of [14C]HMPL-306（Isocitrate Dehydrogenase Inhibitor） in Healthy Chinese Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-306-00CH1
Record Dates: First submitted 2024-10-29; First posted 2024-11-04 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mass Balance Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 100 µCi [14C] HMPL-306 (Experimental): After an overnight fasting of at least 10 hours, subjects will receive [14C] HMPL-306 containing 250 mg HMPL-306 (approximately 100 μCi radioactivity) 30 minutes after start of breakfast (must be completed within 30 minutes) and ensure that all of the drug is taken within 10 minutes.
  Interventions: Drug: 100 µCi [14C] HMPL-306

INTERVENTIONS:
Drug: 100 µCi [14C] HMPL-306 — D1: 250 mg/100 µCi [14C] HMPL-306 Single dose
  Other Names: 100 µCi [14C] HMPL-306 suspension

SUMMARY:
To evaluate the absorption, metabolism and excretion in healthy Chinese male subjects after a single oral dose of [14C]HMPL-306

DETAILED DESCRIPTION:
* To quantitatively analyze the total radioactivity in excreta after oral administration of [14C]HMPL-306 in healthy subjects, obtain the data on human radioactivity excretion rate and determine the main excretion pathways;
* To obtain the radioactive metabolite profile in plasma, urine, and feces after oral administration of [14C]HMPL-306 in healthy subjects, to identify the main metabolites and to determine the metabolism and elimination pathways;
* To quantitatively analyze the total radioactivity in whole blood and plasma in healthy subjects after oral administration of [14C]HMPL-306, to obtain the pharmacokinetics of total radioactivity in plasma and to investigate the distribution of total radioactivity in whole blood and plasma;

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are fully informed about the contents, procedures and possible adverse reactions of the study, voluntarily sign the informed consent form, and are able to communicate well with investigators and to complete all study procedures specified in the protocol;
2. Healthy male subjects who are 18 to 45 years (inclusive) at the time of signing the informed consent form.;
3. Weight ≥50 kg, and body mass index (BMI) between 19 - 26 kg/m2 (inclusive);
4. Subjects must promise to have no pregnancy plan or sperm donation plan and to use condoms during sexual intercourse from signing the informed consent form until 180 days after end of the study treatment. If the sexual partner is a female of childbearing potential, a highly effective method of contraception should be also used (see Appendix 1 for more information).

Exclusion Criteria:

1. History of serious allergy (e.g., drug allergy) and acute allergic rhinitis or food allergy within two weeks prior to screening;
2. Subjects with a history or clinical manifestation of clinically significant metabolic/endocrine, hepatic, renal, hematologic, pulmonary, immunologic, cardiovascular, gastrointestinal, genitourinary, neurologic, or psychiatric diseases within 3 months prior to and during the screening period (judged by investigators);
3. Previous history of hypertension;
4. Subjects who are positive for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibody, anti-human immunodeficiency virus (HIV) antibody, or anti-treponema pallidum antibody;
5. Smoking more than 10 cigarettes daily within 3 months prior to the screening and inability to refrain from smoking completely during the study period;
6. Regular alcohol consumption within 6 months prior to the study, i.e., drinking more than 14 units of alcohol per week (1 unit =360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine), or positive alcohol breath at screening;
7. Presence of drug abuse or dependence, or positive urine screen for drugs of abuse;
8. Subjects who have poor venous access, and have a fear of needles, hemophobia or difficulty in blood collection;
9. Having participated in clinical trials for other drugs within 3 months prior to the screening;
10. Workers who need to be exposed to radioactive condition for a long term; or those who have significant radiation exposure (≥2 times of chest/abdominal computerised tomography (CT), or ≥3 times of other kinds of X-ray examinations) within 1 year prior to administration, or have participated in the radiopharmaceutical labeling study;
11. Subjects who have been vaccinated within 30 days prior to administration and who have a plan for vaccination within 2 weeks after administration;
12. According to the investigator's judgment, the subjects have any other disease or status that may affect the normal completion of the study or the evaluation of the study data, or have any other condition that is not suitable for the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Human Mass Balance | Day1~Day29
  Recovery and cumulative recovery of total radioactivity in excreta (urine and feces).
Human Mass Balance | Day-1~Day29
  Percentage of the unchanged drug and its metabolites in plasma to total radioactivity exposure levels in plasma;
Human Mass Balance | Day-1~Day29
  Percentage of the unchanged drug and its metabolites in urine and feces to the administered dose;
Human Mass Balance | Day-1~Day29
  Identification of major metabolites in plasma, urine and feces.
Human Mass Balance | Day-1~Day29
  PK parameters of total radioactivity in the plasma; Ratio of total radioactivity concentration in whole blood/plasma at different time points.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, offices director, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital)
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR